CLINICAL TRIAL: NCT00246727
Title: Study 1: Effects of a Dietary Supplement (SV) on Advanced NSCLC Treated With Chemotherapy: A Randomized Double Blind Placebo Controlled Study; Study 2: Effects of a Dietary Supplement (SV) on Advanced NSCLC Treated With Best Supportive Care: A Randomized Double Blind Placebo Controlled Study
Brief Title: Effects of Selected Vegetable and Herb Mix (SV) on Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Farm Corporation (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: SV-001 and SV-002; NCT00352274 (obsolete NCT alias); NCT00392626 (obsolete NCT alias)
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study 1: Chemotherapy plus SV or Placebo (Placebo Comparator): For newly diagnosed patients who will be receiving or have received less than 4 weeks of a standard chemotherapy regimen.
  Interventions: Drug: Selected Vegetable and Herb Mix
- Study 2: SV vs Placebo without chemotherapy (Placebo Comparator): For those who have stopped or refuse standard chemotherapy but will receive best supportive care.
  Interventions: Drug: Selected Vegetable and Herb Mix

INTERVENTIONS:
Drug: Selected Vegetable and Herb Mix — The phytomix consists of 19 vegetable and herbs in a highly concentrated form. These vegetables and herbs were selected based on their anti-cancer and immune-enhancing activities. Each batch of raw materials has gone through a very strict quality control (QC) scheme to make sure the product meets our QC standards and devoid of deleterious contaminations, such as heavy metals, pesticides, aflatoxin, and microorganisms. The manufacturing process is tightly controlled to ensure batch-to-batch consistency. The final product, a 20 gram freeze-dried powder, is sealed in a pouch. In our previous studies, patients who ingested phytomix daily for 17-60 months showed no clinical sign of adverse effect.

SUMMARY:
The primary objective of these two studies is to test the hypothesis that the daily ingestion of a dietary supplement, Selected Vegetables and Herbs Mix (SV), which consists of non-toxic botanicals containing known anti-cancer and/or immune enhancing components, may prolong the survival time of stage IIIB/IV non-small cell lung cancer (NSCLC) patients. Either SV or placebo will be added to their daily diet in a double-blind randomized fashion, so that there will be 2 chances out of 3 of receiving SV and 1 chance out of 3 of receiving placebo.

* Study 1: For newly diagnosed patients who will be receiving or have received less than 4 weeks of, a standard chemotherapy regimen.
* Study 2: For those who have stopped or refuse standard chemotherapy but will receive best supportive care.

DETAILED DESCRIPTION:
Carcinoma of the lung is the leading cause of cancer related deaths in North America. Non-small Cell Lung Cancer (NSCLC) causes the death of more than 400,000 patients annually in the US and Western Europe. The benefit of conventional therapies, such as chemotherapy and radiotherapy, for unresectable stage IIIB and IV NSCLC patients is small; the generally accepted median survival time of late stage patients has remained 4-6 months in the "Supportive Care" group and 6-9 months in the chemotherapy treatment group; the one-year survival is about 20%. Ideal Treatment for NSCLC: The toxicity of chemotherapy and side-effects of radiotherapy to the quality of life of the patients have been a major issue in cancer treatments. It has been significant enough that many patients choose to forgo standard treatments. Furthermore, the current chemotherapy for advanced NSCLC is quite expensive, about $50,000 to $100,000 per year. Therefore, an ideal treatment for advanced NSCLC patients should meet the following criteria:

1. Prolong patient survival.
2. Minimal toxicity.
3. Improvement in the patient's quality of life.
4. Relatively inexpensive. A phytomix consisting of selected vegetables and herbs appears to meet all these criteria. The phytomix consists of 19 vegetable and herbs in a highly concentrated form. These vegetables and herbs were selected based on their anti-cancer and immune-enhancing activities. Each batch of raw materials has gone through a very strict quality control (QC) scheme to make sure the product meets our QC standards and devoid of deleterious contaminations, such as heavy metals, pesticides, aflatoxin, and microorganisms. The manufacturing process is tightly controlled to ensure batch-to-batch consistency. The final product, a 20 gram freeze-dried powder, is sealed in a pouch. In our previous studies, patients who ingested phytomix daily for 17-60 months showed no clinical sign of adverse effect.

The Objectives of the proposed studies are to evaluate the benefits and adverse reactions of adding SV to the daily diet of cancer patients who are willing to undergo the chemotherapy (Study 1) or those who refuse chemotherapy (Study 2).

ELIGIBILITY:
Inclusion Criteria:

* Pathological and radiographic documented stage IIIB/IV NSCLC (squamous, adenocarcinoma, bronchioloalveolar, large cell, undifferentiated or not otherwise specified non-small cell carcinoma) diagnosed less than two months prior to randomization. Patients must have ECOG performance status of 0-1 and life expectancy >3 months.
* Patients must never have been diagnosed with any malignancy other than the current NSCLC, except for non-metastatic non-melanoma skin cancer, or cancer in situ of the cervix.
* Patients must be >18 years of age.
* Patients must demonstrate the ability and willingness to eat solid food and SV/placebo.
* Patients must demonstrate the ability and willingness to give informed consent.
* Patients must demonstrate the ability and willingness to follow the study requirements.

Exclusion Criteria:

* Laboratory criteria for exclusion within 14 days prior to randomization.

  * Liver function: bilirubin > 1.5x upper limit of normal (ULN) and SGOT (AST) > 2.5x ULN.
  * Renal function: Serum creatinine >1.5x ULN
  * Bone marrow function: white blood cell (WBC) < 4,000/µl; platelet count < 100,000 mm3; neutrophil count < 1,500/mm3.
  * Hemoglobin <9 gm/dl for males; < 8.5 gm/dl for females.
* Unexplained temperature > 38.5° C for any 7 consecutive days or chronic diarrhea defined as > 3 stools/day persisting for 15 consecutive days, within the 30 days prior to randomization.
* Prior chemotherapy within 5 years.
* Prior radiation to the area of measurable or active tumor.
* Significant cardiac disease (i.e. uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the previous year) or serious cardiac arrhythmia requiring medication.
* Evidence of clinically significant neuropathy (> Grade 1) by physical exam.
* Patients must not be pregnant or breast-feeding. Female patients of child-bearing potential must have a negative pregnancy test performed within 72 hours prior to randomization. Women of child-bearing potential must agree not to become pregnant while participating in the study.
* Active acute infection, except for Herpes viruses (cytomegalovirus [CMV], Epstein Barr virus [EBV], herpes zoster virus [HZV], herpes simplex virus 1 [HSV 1]).
* A serious underlying medical condition other than NSCLC such that life expectancy is less than 2 years.
* Psychiatric illness that may affect the patient's compliance with the treatment.
* Current use of illicit drugs, glucocorticoids other than those necessary for concurrent radiotherapy, adrenal failure or septic shock, or other immune-suppressing or immune-modulating drugs. Glucocorticoids for anti-emetic prophylaxis and therapy should only be used as a last resort.
* A known allergy to one or more components of SV, namely soy beans, mushrooms, mung beans, red dates, scallion, garlic, lentil beans, leek, hawthorn fruit, onions, ginseng, angelica root, Chinese licorice, dandelion root, Senegal root, ginger, olives, sesame seed and parsley.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-12; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Survival Time | Median Survival Time (MST)

SECONDARY OUTCOMES:
Tumor response | After one month of treatment
Quality of Life | For length of study while on active treatment
Toxicity of SV | Annually
  Assessed anually at Safety Monitoring Board

CONTACTS AND LOCATIONS:
Overall Officials: Henry S Sacks, MD, Ph.D, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States